CLINICAL TRIAL: NCT02569801
Title: A Phase II, Open-Label, Randomized Study of GDC-0810 Versus Fulvestrant in Postmenopausal Women With Advanced or Metastatic ER+ /HER2- Breast Cancer Resistant to Aromatase Inhibitor Therapy
Brief Title: A Study of GDC-0810 Versus Fulvestrant in Postmenopausal Women With Advanced or Metastatic Breast Cancer Resistant to Aromatase Inhibitor (AI) Therapy
Acronym: HydranGea
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The Sponsor decided to halt the development of GDC-0810, but not due to any safety concerns.
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GO29689; 2015-000106-19 (EudraCT Number)
Record Dates: First submitted 2015-10-06; First posted 2015-10-07 (Estimated); Results first posted 2021-04-23 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Fulvestrant; 3-(4-(2-(2-chloro-4-fluorophenyl)-1-(1H-indazol-5-yl)but-1-en-1-yl)phenyl)acrylic acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Fulvestrant (Active Comparator): Participants will receive 500 milligrams (mg) of fulvestrant as two intramuscular injections (250 mg each) on Day 1 and Day 15 of Cycle 1, and on Day 1 of each subsequent 28-day cycle until disease progression, unmanageable toxicity, withdrawal of consent, exhaustion of GDC-0810 drug supply, or termination of study by the Sponsor.
  Interventions: Drug: Fulvestrant
- GDC-0810 (Experimental): Participants will receive three 200 mg tablets (total dose = 600 mg) of GDC-0810 orally once daily until disease progression, unmanageable toxicity, withdrawal of consent, exhaustion of GDC-0810 drug supply, or termination of study by the Sponsor.
  Interventions: Drug: GDC-0810

INTERVENTIONS:
Drug: Fulvestrant — Fulvestrant at a dose of 500 mg as two intramuscular injections will be administered on Day 1 and Day 15 of Cycle 1, and on Day 1 of each subsequent 28-day cycle.
  Arms: Fulvestrant
Drug: GDC-0810 — GDC-0810 will be administered as tablets at a dose of 600 mg orally once daily.
  Other Names: RO7056118
  Arms: GDC-0810

SUMMARY:
The primary purpose of this study is to evaluate the efficacy, safety, and tolerability of GDC-0810 compared with fulvestrant in postmenopausal women with advanced or metastatic estrogen receptor positive (ER+)/ human epidermal growth factor receptor 2 negative (HER2-) breast cancer resistant to AI therapy. The development of GDC-0810 has been halted by the Sponsor and the enrollment in this study has been discontinued. Participants currently enrolled in the study who are experiencing clinical benefit may continue receiving GDC-0810 as a single agent or fulvestrant until disease progression (PD), unmanageable toxicity, withdrawal of consent, exhaustion of GDC-0810 drug supply, or termination of the study by the Sponsor.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women with histologically or cytologically confirmed invasive, ER+/HER- (defined by local guidelines) metastatic or inoperable, locally advance breast cancer
* Participants for whom endocrine therapy is recommended and treatment with cytotoxic chemotherapy is not indicated at time of entry into the study
* Participants must have measurable disease by RECIST v1.1 or non-measurable, evaluable disease with atleast one evaluable bone lesion by RECIST v1.1 based on radiologic scans within 28 days of Day 1 of Cycle 1
* Participants with radiologic/objective evidence of breast cancer recurrence or progression while on or within 6 months after the end of adjuvant treatment with an AI, or progression while on or within 1 month after the end of prior AI treatment for locally advanced or metastatic breast cancer

Exclusion Criteria:

* HER2-positive disease
* Prior treatment with fulvestrant
* Prior treatment with greater than (>) 1 cytotoxic chemotherapy regimen or >2 endocrine therapies for advanced or metastatic disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2015-12-04 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (44):
- United States (7):
  - Yale Cancer Center, New Haven, Connecticut
  - Florida Cancer Specialists-Broadway, Fort Myers, Fort Myers, Florida
  - Florida Cancer Specialists (St. Petersburg - St. Anthony's Professional Building), St. Petersburg, Florida
  - Oncology Hematology Care Inc, Cincinnati, Ohio
  - Tennessee Oncology PLLC, Franklin, Tennessee
  - The Center for Cancer and Blood Disorders - Fort Worth, Fort Worth, Texas
  - MD Anderson Cancer Center, Houston, Texas
- Australia (7):
  - St Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - Port Macquarie Base Hospital, Port Macquarie, New South Wales
  - Adelaide Cancer Centre, Kurralta Park, South Australia
  - Royal Hobart Hospital; Medical Oncology, Hobart, Tasmania
  - Footscray Hospital, Footscray, Victoria
  - Peninsula and South Eastern Haematology and Oncology Group, Frankston, Victoria
  - Epworth HealthCare; Clinical Trials Centre, Richmond, Victoria
- Germany (7):
  - Universitätsklinikum "Carl Gustav Carus" der Technischen Universität Dresden, Dresden
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Praxisklinik für Hämatologie und Onkologie Dres. Köppler/Heymans/Weide/Thomalla, Koblenz
  - HELIOS Klinikum Krefeld; Klinik für Frauenheilkunde und Geburtshilfe, Krefeld
  - Rotkreuzklinikum München; Frauenklinik, München
  - Universitätsklinikum Tübingen, Tübingen
  - Marien Hospital Witten Gemeinnützige GmbH, Witten
- South Korea (6):
  - Kyungpook National University Medical Center, Daegu
  - National Cancer Center, Goyang-si
  - Samsung Medical Center, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Korea University Guro Hospital, Seoul
  - Ulsan University Hosiptal, Ulsan
- Spain (10):
  - Hospital Clinic, Barcelona, Cantabria
  - Complejo Hospitalario Universitario A Coruña; Servicio de Endocrinologia, A Coruña, LA Coruña
  - Hospital Universitari Arnau de Vilanova, Lleida, Lerida
  - Hospital del Mar, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hosp. Clinico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Clinico Universitario de Valencia, Valencia
- United Kingdom (7):
  - Royal Sussex County Hospital, Brighton
  - Western General Hospital, Edinburgh
  - St Bartholomew's Hospital, London
  - University College Hospital, London
  - Sarah Cannon Research Institute, London
  - Macclesfield District General Hospital, Macclesfield
  - Nottingham City Hospital, Nottingham

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | GDC-0810 | Fulvestrant
Started (Started=Randomized) | 36 | 35
Received Treatment | 35 | 35
Completed | 0 | 0
Not Completed | 36 | 35
Not completed — Withdrawal by Subject | 9 | 9
Not completed — Sponsor Decision | 13 | 14
Not completed — Progressive Disease | 2 | 7
Not completed — Lost to Follow-up | 0 | 1
Not completed — Death | 12 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GDC-0810 | Fulvestrant | Total
Number analyzed (Participants) | 36 | 35 | 71
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.2 (12.9) | 64.2 (10.5) | 63.2 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 35 | 71
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 13 | 15 | 28
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 22 | 18 | 40
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) in Intent-to-Treat (ITT) Population
Description: PFS was defined as the time from randomization to the first occurrence of disease progression, as determined by investigator review of tumor assessments using RECIST v1.1 or death on study from any cause.
Time Frame: From Day 1 to PD or death from any cause, assessed up to end of study (up to approximately 25 months)
Population: Outcome Measures not assessed based on pre-specified thresholds not having been met.
Arm/Group | GDC-0810 | Fulvestrant
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: PFS According to RECIST v1.1 in Participants With Estrogen Receptor (ESR)1 Mutations
Description: as for outcome 1
Time Frame: From Day 1 to PD or death from any cause, assessed up to end of study (up to approximately 25 months)
Population: Outcome Measures not assessed based on pre-specified thresholds not having been met.
Arm/Group | GDC-0810 | Fulvestrant
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from randomization to death from any cause.
Time Frame: From Day 1 to death from any cause, assessed up to end of study (up to approximately 25 months)
Population: Outcome Measures not assessed based on pre-specified thresholds not having been met.
Arm/Group | GDC-0810 | Fulvestrant
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Percentage of Participants With Objective Response (Partial Response [PR] Plus Complete Response [CR]) According to RECIST v1.1
Description: Objective Response was defined as the percentage of participants who attained CR or PR. CR: Disappearance of all target lesions and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm, PR: At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters.
Time Frame: From Day 1 to PD or death from any cause, assessed up to end of study (up to approximately 25 months)
Measure: Number (90% Confidence Interval); unit: percentage
Arm/Group | GDC-0810 | Fulvestrant
Number analyzed (Participants) | 36 | 35
percentage | 0 [0 to 0] | 8.6 [3.19 to 19.28]

5. Secondary Outcome: Duration of Response (DOR) Assessed Using RECIST v1.1
Description: DOR was defined as the time from first observation of an objective response until first observation of disease progression as assessed by the investigator according to RECIST v1.1 or death from any cause.
Time Frame: From objective response to PD or death from any cause, assessed up to end of study (up to approximately 25 months)
Population: Outcome Measures not assessed based on pre-specified thresholds not having been met.
Arm/Group | GDC-0810 | Fulvestrant
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Percentage of Participants With Clinical Benefit (PR, CR, or Stable Disease, Lasting for At Least 24 Weeks) Assessed Using RECIST v1.1
Time Frame: From Day 1 to PD or death from any cause, assessed up to end of study (up to approximately 25 months)
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | GDC-0810 | Fulvestrant
Number analyzed (Participants) | 36 | 35
percentage of participants | 16.7 [7.52 to 30.22] | 31.4 [19.28 to 44.84]

7. Secondary Outcome: Percentage of Participants With Adverse Events (AEs) and Serious AEs (SAEs)
Time Frame: From Day 1 to 28 days after last dose of study drug, assessed up to end of study (up to approximately 25 months)
Population: Participants who received at least one dose of any study drug
Measure: Number; unit: percentage of participants
Arm/Group | GDC-0810 | Fulvestrant
Number analyzed (Participants) | 35 | 35
percentage of participants
  AEs | 97.1 | 91.4
  SAEs | 20.0 | 14.3

8. Secondary Outcome: GDC-0810 Plasma Concentrations by Visit
Description: Concentration of GDC-0810 measured in plasma after a single dose (Cycle 1 Day 1) and at steady state (Cycle 3 Day 1)
Time Frame: Predose (within 30 minutes of GDC-0810 administration) and 3 hours postdose on Day 1 of Cycles 1 and 3; Cycle length=28 days
Population: Participants who received at least one dose of any study drug and provided a post-dose blood sample in the GDC-0810 arm
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter (ng/mL)
Arm/Group | GDC-0810
Number analyzed (Participants) | 32
Nanograms per milliliter (ng/mL)
  Cycle 1, Day 1 (3 hours post-dose) | 6510 (574)
  Cycle 3, Day 1 (pre-dose): number analyzed (Participants) | 16
  Cycle 3, Day 1 (pre-dose) | 528 (266)
  Cycle 3, Day 1 (3 hours post-dose): number analyzed (Participants) | 15
  Cycle 3, Day 1 (3 hours post-dose) | 10100 (132)

ADVERSE EVENTS:
Time Frame: Up to approximately 25 months
Arm/Group | GDC-0810 | Fulvestrant
All-Cause Mortality (participants affected / at risk) | 12/35 | 4/35
Serious Adverse Events (participants affected / at risk) | 7/35 | 5/35
Other Adverse Events (participants affected / at risk) | 33/35 | 31/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GDC-0810 (N=35) | Fulvestrant (N=35)
CARDIAC TAMPONADE (Cardiac disorders) | 0 (0) | 1 (1)
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1) | 0 (0)
GASTRITIS HAEMORRHAGIC (Gastrointestinal disorders) | 1 (1) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 1 (1) | 0 (0)
BRONCHITIS (Infections and infestations) | 0 (0) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0)
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
BRACHIAL PLEXOPATHY (Nervous system disorders) | 0 (0) | 1 (1)
URINARY TRACT OBSTRUCTION (Renal and urinary disorders) | 1 (1) | 0 (0)
ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 (1) | 0 (0)
LYMPHOEDEMA (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GDC-0810 (N=35) | Fulvestrant (N=35)
ANAEMIA (Blood and lymphatic system disorders) | 3 (4) | 2 (2)
PALPITATIONS (Cardiac disorders) | 1 (1) | 2 (2)
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 3 (3) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 (2) | 1 (1)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 2 (2) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 8 (8) | 6 (7)
DIARRHOEA (Gastrointestinal disorders) | 15 (24) | 8 (10)
DRY MOUTH (Gastrointestinal disorders) | 2 (2) | 1 (1)
DYSPEPSIA (Gastrointestinal disorders) | 4 (4) | 2 (2)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 2 (2) | 2 (2)
NAUSEA (Gastrointestinal disorders) | 11 (12) | 5 (7)
VOMITING (Gastrointestinal disorders) | 10 (14) | 3 (3)
ASTHENIA (General disorders) | 8 (10) | 2 (2)
FATIGUE (General disorders) | 7 (7) | 10 (10)
INJECTION SITE PAIN (General disorders) | 0 (0) | 4 (5)
PNEUMONIA (Infections and infestations) | 2 (2) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 3 (3) | 4 (4)
URINARY TRACT INFECTION (Infections and infestations) | 3 (3) | 2 (3)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 2 (2) | 0 (0)
WEIGHT DECREASED (Investigations) | 1 (1) | 3 (3)
DECREASED APPETITE (Metabolism and nutrition disorders) | 6 (7) | 6 (7)
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 3 (4) | 0 (0)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (4)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 3 (5) | 7 (7)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
MUSCULOSKELETAL STIFFNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
BALANCE DISORDER (Nervous system disorders) | 0 (0) | 2 (2)
DISTURBANCE IN ATTENTION (Nervous system disorders) | 0 (0) | 2 (2)
DIZZINESS (Nervous system disorders) | 3 (3) | 2 (2)
DYSGEUSIA (Nervous system disorders) | 4 (4) | 0 (0)
HEADACHE (Nervous system disorders) | 1 (2) | 3 (3)
ANXIETY (Psychiatric disorders) | 0 (0) | 2 (2)
INSOMNIA (Psychiatric disorders) | 2 (2) | 4 (4)
POLLAKIURIA (Renal and urinary disorders) | 0 (0) | 2 (2)
BREAST PAIN (Reproductive system and breast disorders) | 2 (3) | 0 (0)
VAGINAL DISCHARGE (Reproductive system and breast disorders) | 2 (2) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 6 (7)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
ALOPECIA (Skin and subcutaneous tissue disorders) | 1 (1) | 6 (6)
HOT FLUSH (Vascular disorders) | 0 (0) | 2 (2)
HYPERTENSION (Vascular disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-24): https://cdn.clinicaltrials.gov/large-docs/01/NCT02569801/Prot_SAP_000.pdf